CLINICAL TRIAL: NCT02731963
Title: Mechanical Bowel Preparation for Elective Colorectal Anastomosis: Randomized Clinical Trial.
Brief Title: Mechanical Bowel Preparation for Elective Colorectal Anastomosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CLOTILDE FUENTES OROZCO, PhD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F-2015 1301-18
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Anastomosis
Keywords: Outcomes; Bowel preparation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mechanical bowel preparation (Experimental): 80 Patients who received mechanical bowel preparation with 4 packets of polyethylene glycol in 4 liters of water, 4 hours before intervention.
  Interventions: Drug: Polyethylene glycol
- No mechanical bowel preparation (No Intervention): 81 Patients who received clear liquid diet 1 day before intervention.

INTERVENTIONS:
Drug: Polyethylene glycol — Patients with colorectal pathology who underwent elective colorectal anastomosis, that were randomized into two groups; one of them received mechanical bowel preparation with polyethylene glycol (study group), and the other one received clear liquid diet(control group) .
  Arms: Mechanical bowel preparation

SUMMARY:
Colorectal surgery is highly associated with septic complications, therefore, multiple approaches have been used to reduce this complications, one of the most used is mechanical bowel preparation. Lately multiple studies have suggested that mechanical bowel preparation might not be necessary.

DETAILED DESCRIPTION:
Objective: Compare elective colorectal anastomosis with or without mechanical bowel preparation on outcomes, particularly anastomotic leak, surgical site infection, and ileum.

Materials and methods: A clinical trial was conducted including patients with colorectal pathology who underwent elective colorectal anastomosis. Patients were randomized into two groups; with mechanical bowel preparation (Group 1), and without mechanical bowel preparation (Group 2). Surgical, and non-surgical outcomes were evaluated, including anastomotic leak, surgical site infection, ileum, acute kidney injury, pneumonia, and mortality.

The statistical analysis was performed according to the nature of variables, for continuous data using measures of central tendency and dispersion and for the qualitative data with frequencies and percentages. Inferential analysis with student's t-test, and/or Mann-Whitney's U test; chi-square distribution, and/or Fisher's exact test respectively.

ELIGIBILITY:
Inclusion Criteria:

* Entitlement to the Mexican Institute of Social Security
* Signed informed consent
* Patients with colorectal pathology who needed primary elective colorectal anastomosis
* Body mass index >18, and < 31

Exclusion Criteria:

* Patients who dropped out from the study or withdrew the informed consent
* Patients who did not accepted the surgical procedure
* Patients who had been submitted to surgery before entering the protocol
* Patients who need a colostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Anastomotic leak | 6 weeks
  Following the surgical procedure, anastomotic leak was evaluated with fecal discharge on drainage and confirmed with computerized tomography.
Number of Participants with Surgical site infection | 6 weeks
  Following the surgical procedure, surgical site infection was evaluated if the patient presented specific signs and symptoms for this condition (redness, delayed healing, fever, pain, tenderness, warmth, or swelling), and confirmation with culture of the purulent discharge.
Number of Participants with Postoperative ileus | 6 weeks
  Following the surgical procedure, ileus was evaluated if the patient presented distended and tympanic abdomen, and absence or hypoactive bowel sounds, and confirmed with a plain abdominal radiography.

SECONDARY OUTCOMES:
Number of Participants with Fistula | 6 weeks
  Following the surgical procedure, fistula was evaluated with fecal discharge on drainage and confirmed with CT fistulography.
Number of Participants with Abdominal sepsis | 6 weeks
  Following the surgical procedure, abdominal sepsis was evaluated if the patient presented specific signs and symptoms for this condition (fever, abdominal pain, ascites, worsening), and confirmation with computerized tomography.
Number of Participants with Abscess | 6 weeks
  Following the surgical procedure, abscesses were evaluated if the patient presented specific signs and symptoms for this condition (fever, abdominal pain, ascites), and confirmation with computerized tomography.
Number of Participants with Pneumonia | 6 weeks
  Following the surgical procedure, pneumonia was evaluated if the patient presented specific signs and symptoms for this condition (fever, shaking chills, cough productive of sputum), and confirmation with chest radiography.
Number of Participants with Acute kidney injury | 6 weeks
  Following the surgical procedure, acute kidney injury was evaluated with kidney function studies (BUN, creatinine)

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided